CLINICAL TRIAL: NCT04940897
Title: Use of Capillary Blood Ketone Meters to Improve Ambulance Service Care of Hyperglycaemic Patients: a Feasibility Study
Brief Title: Use of Blood Ketone Meters to Improve Ambulance Hyperglycaemia Care
Acronym: KARMA2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East of England Ambulance Service NHS Trust (Other Government)
Responsible Party: Principal Investigator, Theresa Foster, Head of Research, East of England Ambulance Service NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KARMA2
Record Dates: First submitted 2021-05-25; First posted 2021-06-28 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Diabetic Ketoacidosis
MeSH Terms: conditions — Diabetic Ketoacidosis

STUDY DESIGN:
Intervention Model Description: Stepped wedge control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Usual care plus ketone meter and fluid therapy for identified high risk DKA patients
  Interventions: Other: Use of CareSens ketone meter

INTERVENTIONS:
Other: Use of CareSens ketone meter — Use of CareSens ketone meter to identify blood ketone levels and delivery of fluid therapy to those patients at high risk of DKA

SUMMARY:
In this KARMA2 feasibility study the investigators are testing whether ambulance staff can reliably and safely identify patients at high risk of diabetic ketoacidosis using blood ketone meters and start fluid (saline) therapy before arriving at hospital. The investigators aim to include 800 patients in this stepped wedge control study and the results will help decide if a larger study is warranted.

DETAILED DESCRIPTION:
Diabetic ketoacidosis (DKA) is a potentially life-threatening condition which requires immediate treatment. National Health Service (NHS) hospital guidelines recommend immediate fluid (saline) therapy. Delays in diagnosis and treatment are known to be associated with health complications and death.

There is an opportunity to involve ambulance crews to improve DKA identification and treatment times; however, currently ambulance staff do not have access to ketone testing, and fluids are recommended only when it is thought a patient is critically unwell.

In this KARMA2 feasibility study the investigators are testing whether ambulance staff can reliably and safely identify patients at high risk of DKA using blood ketone meters and start fluid (saline) therapy before arriving at hospital.

During an 8-month period (4-month control followed by 4-month intervention), 120 ambulance clinicians from the East of England Ambulance Service NHS Trust will receive training to consent 400 patients with hyperglycaemia and unwell patients with diabetes to the control group receiving usual care, followed by determining the presence of ketones using capillary blood testing from a further 400 consenting patients with hyperglycaemia and unwell patients with diabetes. Subsequent patient care will depend on the ketone value obtained: high-risk DKA patients will receive fluid therapy.

Twenty ambulance and hospital clinicians will be invited to an online interview to share views of DKA care and the impact of ambulance blood ketone meters. The results will help the investigators decide if a larger study would be a good idea.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or more
* Attended by study clinician
* Informed or Proxy consent to participate
* Blood glucose level greater than 11mmol/L or unwell with history of diabetes
* If required will be transported to partner hospital

Exclusion Criteria:

* Failure to meet inclusion criteria
* Previously recruited to study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Measure incidence of hyperglycaemia in study population | 18 months
  Frequency count of capillary blood glucose level greater than 11mmol/L
Measure incidence of diabetic ketoacidosis (DKA) in study population | 18 months
  Frequency count of capillary blood ketone level equal to or greater than 3mmol/L
Completeness of data capture by study clinicians | 18 months
  Progression criteria requires full record completion for a minimum of 70 percent of participants
Measure incidence of adverse events | Maximum 18 months
  Progression criteria requires adverse event rate to be less than 1 percent of participants

CONTACTS AND LOCATIONS:
Overall Officials: Tom Davis, Study Director — East of England Ambulance Service NHS Trust
Locations (1):
- East of England Ambulance Service NHS Trust, Melbourn, Cambs, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prothero LS, Strudwick T, Foster T, Lake AK, Boyle A, Clark A, Williams J, Rayman G, Dhatariya K. Ambulance clinician use of capillary blood ketone meters to improve emergency hyperglycaemia care: A stepped-wedged controlled, mixed-methods feasibility study. Diabet Med. 2024 Sep;41(9):e15372. doi: 10.1111/dme.15372. Epub 2024 Jun 9. PMID 38853420